CLINICAL TRIAL: NCT05321563
Title: Evaluating the Effectiveness of a Drug Education and Diversion Program for Middle and High School Students
Acronym: iDECIDE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to changes in state policy, the need for a comprehensive Tier 2 diversion program became apparent. The PI and Project Officer at MA DPH opened up programming statewide and updated the evaluation plan (NCT06115746).
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Department of Health (Other Government)
Responsible Party: Principal Investigator, Randi Melissa Schuster, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021P002611; INTF2300H78500224179 (Other Grant/Funding Number: Massachusetts Department of Public Health); INTF2400H78500224455 (Other Grant/Funding Number: Massachusetts Department of Public Health)
Record Dates: First submitted 2022-03-18; First posted 2022-04-11 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Adolescent Behavior; Substance Use; Youth; Health Risk Behaviors
Keywords: Diversion Program; Adolescent Substance Use; Middle and High School Students; Indicated Early Intervention; Tier 2 Services; School-Based Intervention
MeSH Terms: conditions — Adolescent Behavior; Substance-Related Disorders; Health Risk Behaviors

STUDY DESIGN:
Intervention Model Description: This is a type 1, hybrid effectiveness-implementation trial using a stepped wedge design with stratified, clustered randomization. Investigators will randomly allocate the timing of implementation of the iDECIDE curriculum compared to standard disciplinary response, over approximately 24 months. Schools will cross over from control (i.e., standard disciplinary response) to intervention (i.e., iDECIDE curriculum) with all schools exposed to iDECIDE by the end of the trial.
Who Masked: Outcomes Assessor
Masking Description: Individuals collecting longitudinal student-level data for the primary aims will be blind to group assignment. Initial implementation of analyses for primary aims will also be 'analyst-blind.' Analyses for primary aims will first be implemented on data where the key factor of interest (whether the 45-day and 90-day follow-ups occurred post-intervention) has been randomly shuffled. Only once data exclusion criteria have been finalized, models have been properly specified, and any other unforeseen circumstances addressed, will the un-shuffled data be provided to the analyst for the final analysis implementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Observation Phase (No Intervention): Schools will continue to apply their standard disciplinary response to school-based substance use infractions during the 'unexposed' study period.
- Intervention Phase (Experimental): Schools will have the opportunity to deliver the iDECIDE curriculum in lieu of or as part of the standard disciplinary response to school-based substance use infractions during the 'exposed' study period.
  Interventions: Behavioral: iDECIDE (Drug Education Curriculum: Intervention, Diversion, and Empowerment)

INTERVENTIONS:
Behavioral: iDECIDE (Drug Education Curriculum: Intervention, Diversion, and Empowerment) — iDECIDE is a 4 session curriculum that addresses topics such as the neurobiology of substance use, adolescent brain development, industry tactics, motivations for using substances, risk and protective factors, triggers, healthy alternatives, core values, and long-term goal setting. These topics are taught via facilitated discussions, videos, worksheets, and handouts. Facilitators are selected by schools and community agencies to receive free trainings conducted by the iDECIDE team, which includes personnel from the Massachusetts Department of Public Health, Massachusetts General Hospital (MGH) Center for Addiction Medicine, and the Institute for Health and Recovery.
  Arms: Intervention Phase

SUMMARY:
The primary goal of this study is to evaluate the effectiveness of the iDECIDE curriculum as an alternative to punitive responses for school-based substance use infractions.

DETAILED DESCRIPTION:
The primary goal of this study is to evaluate the effectiveness of the iDECIDE curriculum as an alternative to punitive responses for school-based substance use infractions. To accomplish this aim, investigators will conduct a Type 1, hybrid effectiveness-implementation trial. Using a stepped wedge design, investigators will randomly allocate the timing of implementation of the iDECIDE curriculum compared to standard disciplinary response, over approximately 24 months. Investigators are testing the overarching hypothesis that student-level outcomes improve when schools transition from a standard disciplinary response to having access to a more educational and therapeutic alternative. Participants for this aim will include students referred by schools with substance use infractions who are assessed by the study team at baseline (proximal to the time of infraction), 45, and 90 days later.

Exploratory aims of this study include:

1. Change in school environment -- Evaluating the impact of transition from punitive responses for substance use to iDECIDE on overall prevalence of substance use and perceptions of school culture. Participants for this exploratory aim include all students within participating schools (not just those with substance use infractions), assessed annually beginning Fall 2022.
2. Single arm pre/post change -- Evaluating change from session 1 to session 4 of iDECIDE in perceptions of harm from substance use, knowledge of drug effects, perceptions of a supportive school culture, plans to change substance use, and frequency of past 7-day substance use in all students who complete the iDECIDE curriculum. Investigators will also explore whether any change in these outcomes differ among historically underserved populations, including racial and gender minority students. Participants for this exploratory aim incIude all students who participate in the iDECIDE curriculum, regardless of the reason for referral into the program and the provision of parental consent for collection of data for primary aims.
3. Identification of implementation barriers -- Evaluating the feasibility and acceptability of the iDECIDE curriculum by identifying multi-level barriers and facilitators to implementation using mixed methods. Participants for this exploratory aim include school stakeholders, interviewed right before and 6 months following iDECIDE implementation.

ELIGIBILITY:
Eligibility criteria for the primary aim (i.e., evaluating how student-level outcomes change when schools transition from a standard disciplinary response to having access to a more educational and therapeutic alternative):

Inclusion Criteria:

* Enrolled in a participating middle or high school;
* Received a substance use-related infraction at school or school-sanctioned event;
* Have a parent or legal guardian who is able and willing to provide written informed consent (if under the age of 18);
* Competent and willing to provide written informed consent (if age 18+) or assent (if under 18);
* Able to read and write comfortably in English;
* In the opinion of the investigator, able to safely participate in the protocol.

Exclusion Criteria:

* Passive consent for referral to MGH evaluation team declined by parent or legal guardian;
* Gross cognitive impairment, for example due to florid psychosis, intellectual disability, developmental delay, or neurodegenerative disease;
* Ward of the state.

Eligibility criteria for participants for exploratory aims:

In addition to the students with school-based substance use infractions enrolled for the primary aims, three additional cohorts of participants will be recruited for exploratory aims. The eligibility criteria for these cohorts are listed below.

Exploratory Aim 1: evaluating the impact of transition from punitive responses for substance use to iDECIDE on overall prevalence of substance use and perceptions of school culture (Annual School-Wide Assessment)

Inclusion Criteria:

* Currently enrolled in a participating middle or high school;
* Provide informed assent/consent for participation in this research by voluntarily completing the survey.

Exclusion Criteria:

* Passive consent for school-wide assessment declined by parent or legal guardian;
* Not able to adequately read and respond to survey items in one of the languages available.

Exploratory Aim 2: Evaluating change from session 1 to session 4 of iDECIDE in perceptions of harm from substance use, knowledge of drug effects, perceptions of a supportive school culture, plans to change substance use, and frequency of past 7-day substance use in all students who complete the iDECIDE curriculum.

Inclusion Criteria:

* Enrolled in the iDECIDE curriculum by a trained iDECIDE facilitator.

Exclusion Criteria:

* Unable to adequately read and respond to survey items in one of the languages available.

Ages: 10 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Knowledge of drug effects from baseline to 90 day follow-up | Baseline - 90 days
  Knowledge of drug effects will be measured by number of items correct on a survey examining a student's understanding of adolescent brain development, neurobiology of addiction, and the impact of alcohol, cannabis, nicotine and other substance use on the brain and body.
Frequency of substance use from baseline to 90 day follow-up | Baseline - 90 days
  Frequency of substance use will be operationalized as the number of days spent using student's preferred substance assessed via 14-day timeline followback.

SECONDARY OUTCOMES:
Emotional support from baseline to 90 day follow-up | Baseline - 90 days
  Quality of relationships with teachers/administrators, school connectedness, and social and emotional satisfaction at school will be measured using summed scores from the NIH Toolbox Emotional Support Fixed Form Ages 8-17 v2.0, modified to specifically query about emotional support from adults in school. Raw scores range from 7 to 33 (age- and gender- corrected T-scores also available), with higher scores indicative of more social support.

CONTACTS AND LOCATIONS:
Overall Officials: Randi M Schuster, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie reported results (after deidentification [text, tables, figures, and appendices]), and the study protocol, statistical analysis plan, analytic code, and informed consent form will be made available to researchers who provide a methodologically sound proposal beginning 3 months and ending 5 years following article publication to achieve aims in the approved proposal. Proposals should be directed to rschuster@harvard.mgh.edu. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement.

REFERENCES:
- [Background] Gray CA, Iroegbulem V, Deming B, Butler R, Howell D, Pascale MP, Bodolay A, Potter K, Turncliff A, Lynch S, Whittaker J, Ward J, Maximus D, Pachas GN, Schuster RM. A pragmatic clinical effectiveness trial of a novel alternative to punishment for school-based substance use infractions: study protocol for the iDECIDE curriculum. Front Public Health. 2023 Aug 21;11:1203558. doi: 10.3389/fpubh.2023.1203558. eCollection 2023. PMID 37670822
- See also: Curriculum Webpage — http://www.idecidemyfuture.org